# Statistical Analysis Plan of the 'Driving Pressure During General Anesthesia for Open Abdominal Surgery' trial (DESIGNATION)

NCT: 03884543

The DESIGNATION-investigators

Amsterdam University Medical Centers, location AMC, Amsterdam, The Netherlands:

Department of Intensive Care

Monash University, Melbourne, Australia

Australian and New Zealand Intensive Care Research Centre

Hospital Israelita Albert Einstein; São Paulo, Brazil:
Department of Critical Care Medicine

Mahidol University, Bangkok, Thailand: Mahidol–Oxford Tropical Medicine Research Unit (MORU)

#### **INTRODUCTION**

The 'Driving Pressure During General Anesthesia for Open Abdominal Surgery' randomized clinical trial (DESIGNATION) compares an intraoperative ventilation strategy with individualized high positive end–expiratory pressure (PEEP) with recruitment maneuvers ('individualized high PEEP') to a conventional strategy with standard PEEP of 5 cmH<sub>2</sub>O without recruitment maneuvers ('low PEEP').<sup>1</sup> The primary objective of this study is to determine whether 'individualized high PEEP' is superior to a 'low PEEP' with regard to the incidence of postoperative pulmonary complications (PPC). Enrollment of patients in DESIGNATION already started and the study is planned to finish around the second trimester of 2024.

To prevent outcome reporting bias and data-driven analysis results, the International Conference on Harmonization of Good Clinical Practice (ICH-GCP) recommends that clinical trials should be analyzed according to a pre-specified detailed Statistical Analysis Plan (SAP).

This document presents the updated and finalized SAP of the DESIGNATION trial.

#### **METHODS**

Design, ethics and registration

DESIGNATION is an international, multicenter, parallel, two–group, prospective, randomized, patient and outcome–assessor blinded superiority clinical trial designed to determine if an individualized intra–operative high PEEP strategy guided by the driving pressure ( $\Delta P$ ) is superior to a standard low PEEP strategy with respect to the development of PPC in adult patients that are at risk for PPC and submitted to open abdominal surgery.

The protocol, with a detailed description of the study population, the two strategies and follow–up plan of the DESIGNATION trial was published elsewhere. The DESIGNATION trial was approved by the Institutional Review Board of the Amsterdam University Medical Centers, location Academic Medical Center, in Amsterdam, The Netherlands (2018\_319, February 7, 2019) and is registered with clinicaltrials.gov (NCT03884543).

#### Randomization and blinding

Eligible patients are randomly allocated in a 1:1 ratio to the 'individualized high PEEP' or 'low PEEP' strategy. The allocation sequence is computer–generated by an independent investigator using permuted blocks of different block sizes, with a maximum block size of eight and stratified per center and BMI (≤ 30 vs. > 30 kg/m²). Randomization is performed by local investigators patient–by–patient employing a dedicated, password protected, SSL–encrypted website.

At each site, at least two investigators are involved with the study. One investigator randomizes the patients immediately before surgery and is responsible for the trial intervention and data collection. A second investigator remains blinded for the randomization and is responsible for postoperative data

collection. The surgeon and patient are kept blind to the allocated ventilation strategy. Since PEEP can be adjusted at any time point upon the surgeons' request or because of concerns about patient's safety, and since patients do not profit from knowing to which group they are allocated to, unblinding is not applicable.

#### Outcomes

The primary study outcome is a collapsed composite of PPC developing within the first five postoperative days. This endpoint follows the European Perioperative Clinical Outcome (EPCO) definition and has been used before in several studies.<sup>2-4</sup> Patients who develop a least one complication are considered as meeting the primary outcome. The components of the composite outcome of PPC have been defined elsewhere,1 and these include: 1) severe respiratory failure; 2) bronchospasm; 3) suspected pulmonary infection; 4) new pulmonary infiltrates; 5) aspiration pneumonitis; 6) new atelectasis; 7) acute respiratory distress syndrome (ARDS); 8) new pleural effusion; 9) new cardiopulmonary edema; and 10) new pneumothorax. The selected PPC can sensibly be added together as they share common pathophysiological mechanisms and have plausibility to be affected in the same direction by the intervention to be tested in this study. If pulmonary infiltrates, pleural effusion, atelectasis, cardiopulmonary edema or pneumothorax are already present in any preoperative chest imaging and did not worsen, the patient will not be coded as a new complication in the postoperative period if present.

Secondary outcomes also have been defined elsewhere,<sup>1</sup> and include: 1) mild respiratory failure; 2) a composite outcome of intraoperative complications, including desaturation, hypotension, any need for vasoactive agents, and any

new arrhythmias; 3) postoperative extrapulmonary complications; 4) intraoperative fluid balance; 5) impaired wound healing; 6) unplanned admission to an ICU; 7) length of intensive care unit (ICU) stay (if applicable); 8) length of hospital stay; and 9) all—cause hospital mortality. All definitions are available in **Table 1**.

#### Cleaning and closing of the database

The database will be locked as soon as all data are entered and all discrepant or missing data are resolved, after all efforts are employed to complete the database, and we consider that the remaining issues cannot be fixed. At this step, the data will be reviewed before database locking. After that, the study database will be locked and exported for statistical analysis. At this stage, permission for access to the database will be removed for all investigators, and the database is locked and archived.

#### Missing data

No or minimal losses to follow-up for the primary outcome is anticipated. Complete-case analysis will be carried out for all outcomes. However, if more than 5% of missing data is found for the primary outcome, a sensitivity analysis using multiple imputations and estimating-equation methods will be carried out. Multiple imputation will consider imputation models based on prognostic baseline and post-baseline variables under a missing at random assumption.

#### Sample size

DESIGNATION is designed to enroll a total of 1.468 patients (734 in each arm). This number allows the detection of a reduction in the incidence of the primary outcome from 34% in the control group to 27.2% in the experimental group (relative risk reduction of 20%), considering a type I error of 5%, a power of 80%,

similar allocation ratio between the arms (1:1) and a dropout rate of 2%. The required sample size is calculated based on an estimated effect size derived from individual patient data from previous trials.<sup>3-8</sup>

#### Statistical analyses

All statistical analyses will be conducted on an intention—to—treat basis, with patients analysed according to their assigned treatment arms, except for cases lost to follow up or withdrawal of informed consent. In addition, a per—protocol analysis will be conducted. Variables will be expressed as counts and percentages, means and standard deviations (SD), or medians and interquartile ranges (IQR) whenever appropriate.

The primary and secondary outcomes will be assessed using a two–sided superiority hypothesis test with a significance level of 0.05 and presented with a two–sided 95% confidence interval. In addition to the unadjusted *p* values for secondary outcomes, a Holm–Bonferroni procedure will be applied to control for multiple testing.<sup>9</sup> Analyses will be performed using the software R (R Core Team, 2016, Vienna, Austria). A list of proposed tables and figures is in **Table 2**.

#### Trial profile

Patient flows will be represented in a CONSORT flowchart (Figure 1).

#### Baseline characteristics

A description of the baseline characteristics of the trial participants will be presented by treatment group (**Table 3**). Discrete variables will be summarized as numbers (%). Percentages will be calculated according to the number of trial participants for whom data are available. Where values are missing, the denominator will be stated in the table and no assumptions or imputations will be made. Continuous variables will be summarized by either means and standard

deviations (SD) or medians and interquartile ranges (IQR), according to the observed distribution of the variable.

#### Adherence to study interventions and ventilatory variables

Surgical and perioperative characteristics will be reported (**Tables 4** and **5**). Ventilatory variables and vital signs will be reported after intubation, one hour, and in the last hour of surgery and compared between the two groups. Absolute differences between groups will be calculated using median regression for continuous variables (reported as median difference) and generalized linear models with binomial distribution and an identity link for binary variables (reported as difference in percentages). Plots comparing ventilatory variables and vital signs among the groups during the first three hours of surgery and in the last hour will be constructed (presenting the data as mean and 95% confidence interval in each time point).

#### Other daily characteristics

Daily variables will be reported according to the description in **Table 6**. Absolute differences between groups will be calculated using median regression for continuous variables (reported as median difference) and generalized linear models with binomial distribution and an identity link for binary variables (reported as difference in percentages). Plots comparing daily variables among the groups will be constructed (presenting the data as mean and 95% confidence interval in each time point).

#### Primary outcome

The effect of 'individualized high PEEP' compared to low PEEP of the incidence of PPC will be assessed using a mixed-effect generalized linear model with binomial distribution and identity link, with sites included as random effects to

account for the clustering effect and reported as absolute difference with a two-sided 95% confidence interval. Results will be presented in a table of outcomes (**Table 7**). To support interpretation, a confidence distribution for the primary outcome using a normal approximation on the estimated absolute difference will be calculated.<sup>10</sup> The confidence distribution will be computed to provide the frequentist probability that the absolute difference is less than 0.<sup>10</sup> In addition, the confidence distribution will be reported in a plot.

#### Secondary outcomes

For binary outcomes, the effect of 'individualized high PEEP' compared to 'low PEEP' on the incidence of PPC will be assessed using a mixed–effect generalized linear model with binomial distribution and identity link, with sites included as random effects to account for the clustering effect and reported as absolute difference with a two–sided 95% confidence interval. For continuous outcomes, the comparison will be made using a mixed-effect median regression with sites also including as clustering effect, and reported as median difference with a two–sided 95% confidence interval. In addition, a Holm–Bonferroni correction to control the family–wide error rate to the *p* values for all 17 secondary outcomes will be done and presented in a Table.

#### Per-protocol analysis

The analysis for the primary endpoint will be repeated in patients who received treatment according to their respective randomisation arm. This includes patients with pre-approved protocol deviations. However, patients with non-pre-approved protocol deviations and protocol violations will be excluded.

#### Subgroup analysis

Treatment effects on incidence of PPC will be analyzed according to the following predefined subgroups: 1) age < 65 years  $vs \ge 65$  years; 2) body mass index < 30 kg/m² vs BMI  $\ge 30$  kg/m²; 3) baseline SpO₂ < 96% vs SpO₂  $\ge 96\%$ ; 4) moderate vs high risk for PPC according to the ARISCAT risk score (< 45 vs.  $\ge 45$ ); 5) duration of surgery < 3 hours  $vs \ge 3$  hours; and 6) planned destination to ICU or HDU vs ward. Analyses of heterogeneity of effects across subgroups will be performed with the use of treatment–by–subgroup term added to the primary model and will be presented in a forest plot.

#### Other exploratory analyses

Since the primary outcome of the present study is a composite one, the choice of the statistical method is an important part of designing because various methods provide different power, depending on the situation. In addition to the standard analysis described above, the following analyses will be performed:

- Count analysis: the number of positive component events (i.e., 'count')
  across the composite will be assessed; the groups will be compared on
  the count using a Wilcoxon rank sum test, and the odds ratio with the 95%
  confidence interval will be assessed with a proportional odds logistic
  regression model;
- Individual component analysis: the effect of the intervention in each component will be analyzed estimating the risk ratio and confidence intervals with Wald's likelihood ratio approximation test using a Bonferroni correction for multiple comparisons; the 99.5% Bonferroni—corrected confidence intervals will be reported (1 0.05/10 = 0.995);

- Common effect test: a multivariate (i.e., multiple outcomes per subject)
   generalized estimating equations (GEE) model will be used to estimate a
   common effect odds ratio across the components;
- Average relative effect test: the average relative effect test will be
  assessed by averaging the component-specific treatment effect from the
  distinct effects model, and testing whether the average is equal to zero. In
  the GEE distinct effect model a distinct treatment effect is estimated for
  each component; and
- Heterogeneity of treatment effect: heterogeneity of treatment effect across components will be assessed by a treatment-by-component interaction test in the distinct effects GEE model.

#### **REFERENCES**

- 1. DESIGNATION-investigators. Driving Pressure During General Anesthesia for Open Abdominal Surgery (DESIGNATION): study protocol of a randomized clinical trial. Trials 2020;21:198.
- 2. Jammer I, Wickboldt N, Sander M, et al. Standards for definitions and use of outcome measures for clinical effectiveness research in perioperative medicine: European Perioperative Clinical Outcome (EPCO) definitions: a statement from the ESA-ESICM joint taskforce on perioperative outcome measures. Eur J Anaesthesiol 2015;32:88–105.
- 3. Hemmes SN, Gama de Abreu M, Pelosi P, Schultz M. High versus low positive end-expiratory pressure during general anaesthesia for open abdominal surgery (PROVHILO trial): a multicentre randomised controlled trial. Lancet 2014;384:495–503.
- 4. Ferrando C, Soro M, Unzueta C, et al. Individualised perioperative openlung approach versus standard protective ventilation in abdominal surgery (iPROVE): a randomised controlled trial. Lancet Respir Med 2018;6:193–203.
- 5. Futier E, Constantin JM, Paugam-Burtz C, et al. A trial of intraoperative low-tidal-volume ventilation in abdominal surgery. N Engl J Med 2013;369:428–37.
- 6. Ge Y, Yuan L, Jiang X, Wang X, Xu R, Ma W. Effect of lung protection mechanical ventilation on respiratory function in the elderly undergoing spinal fusion. J Cent South Univ 2013;38:81–5.
- 7. Severgnini P, Selmo G, Lanza C, et al. Protective mechanical ventilation during general anesthesia for open abdominal surgery improves postoperative pulmonary function. Anesthesiology 2013;118:1307–21.

- 8. Ferrando C, Soro M, Unzueta C, et al. Rationale and study design for an individualised perioperative open-lung ventilatory strategy with a high versus conventional inspiratory oxygen fraction (iPROVE-O2) and its effects on surgical site infection: study protocol for a randomised controlled trial. BMJ Open 2017;7:e016765.
- Holm S. A simple sequentially rejective multiple test procedure. Scand J Stat 1979; 6:65-70.
- 10. Marschner IC. Confidence distributions for treatment effects in clinical trials: Posteriors without prior. Stat Med 2024;43:1271-89.

Table 1 - Definitions of Outcomes

| Outcomes | Definition |
|---|---|
| Severe respiratory failure | Need for noninvasive or invasive mechanical ventilation, or a $PaO_2 < 60$ mmHg (or $< 7.9$ kPa) or $SpO_2 < 90\%$ despite supplemental oxygen in spontaneously breathing patients. |
| Bronchospasm | Newly detected expiratory wheezing treated with bronchodilators. |
| Suspected pulmonary infection | <ul> <li>Receiving antibiotics and meeting at least one of the following criteria:</li> <li>New or changed sputum;</li> <li>New or changed lung opacities on chest radiograph when clinically indicated;</li> <li>Tympanic temperature &gt; 38.3 °C;</li> <li>White blood cell count &gt; 12,000/μL.</li> </ul> |
| Pulmonary infiltrates | Any unilateral or bilateral infiltrates on chest radiography. |
| Aspiration pneumonitis | Respiratory failure after the inhalation of regurgitated gastric contents. |
| Atelectasis | Lung opacification with shift of the mediastinum, hilum, or<br>hemidiaphragm towards the affected area, and<br>compensatory overinflation in the adjacent non-<br>atelectasis lung on chest radiography. |
| Acute respiratory distress syndrome | According to the Berlin criteria for acute respiratory distress syndrome*. |
| Pleural effusion | Blunting of the costophrenic angle, loss of the sharp silhouette of the ipsilateral hemidiaphragm in upright position, evidence of displacement of adjacent anatomical structures, or (in supine position) a hazy opacity in one hemithorax with preserved vascular shadows on chest radiography. |
| Cardiopulmonary edema | Clinical signs of congestion, including dyspnea, edema, rales and jugular venous distention, with the chest radiograph demonstrating increase in vascular markings and diffuse alveolar interstitial infiltrates. |
| Pneumothorax | Air in the pleural space with no vascular bed surrounding the visceral pleura on chest radiography. |
| Mild respiratory failure | $PaO_2 < 60$ mmHg (or < 7.9 kPa) or $SpO_2 < 90\%$ in room air, but responding to supplemental oxygen (excluding hypoventilation). |
| Intraoperative desaturation | $SpO_2 \le 90\%$ or if preoperative $SpO_2 < 90\%$ an absolute decrease in $SpO_2 > 5\%$ and lasting > 1 minute. |
| Intraoperative hypotension | Decrease in mean arterial pressure of > 20% and lasting for > 3 minutes. |
| Intraoperative need for vasoactive agents | Vasoactive agents more than needed to compensate for vasodilating effects of anesthesia. |
| Intraoperative arrhythmias | Needing intervention as suggested by the Advanced Cardiac Life Support Guidelines**. |
| Sepsis | According to SEPSIS-3 criteria***. |
| Septic shock | According to SEPSIS-3 criteria***. |
| Extrapulmonary infection | Wound infection plus any other infection. |
| Acute kidney injury | According to Acute Kidney Injury Network (AKIN) criteria**** Detail Acute respiratory distress syndrome: the Berlin Definition, IAMA |

<sup>\*</sup> ARDS Definition Task Force, Ranieri VM, Rubenfeld GD, et al. Acute respiratory distress syndrome: the Berlin Definition. JAMA

<sup>2012;307:2526-33.

\*\*</sup> Link MS, Berkow LC, Kudenchuk PJ, et al. Part 7: Adult Advanced Cardiovascular Life Support: 2015 American Heart Association

\*\*Configuration 2015:132:444-64 Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation 2015;132:444-64. \*\*\* Singer M, Deutschman CS, Seymour CW, et al. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA 2016;315:801–10.

\*\*\*\* Mehta RL, Kellum JA, Shah SV, et al. Acute Kidney Injury Network: report of an initiative to improve outcomes in acute kidney

injury. Crit Care 2007;11:R31.

Table 2 – List of proposed tables and figures

| | Description |
|---|---|
| Main paper | · |
| Table 1 | Baseline Characteristics of the Included Patients |
| Table 2 | Ventilation and Intraoperative Characteristics |
| Table 3 | Primary and Secondary Outcomes |
| Figure 1 | Participant Flow Diagram |
| | Postoperative Pulmonary Complications in Prespecified Subgroups |
| Figure 2 | A forest plot showing the absolute difference and two-sided 95% confidence intervals with p value for interaction calculated via a test for treatment-by-subgroup interaction in |
| Online Cumpl | the regression model. A solid line of reference in the number 1 and a dashed line of reference in the overall effect will be shown. |
| Online Suppl | |
| eTable 1 | Rate of Missing Data A table showing the rate of missing data. |
| | Additional Intraoperative Characteristics |
| eTable 2 | A table showing additional intraoperative characteristics. |
| oToble 2 | Rescue Therapies in Included Patients |
| eTable 3 | A table showing the steps of rescue therapies in patients receiving rescue in each arm. |
| eTable 4 | Protocol Deviations |
| CTUDIO I | A table reporting the protocol deviations in each arm. |
| eTable 5 | Daily Assessment of Included Patients |
| | A table showing characteristics over the first 5 days of follow-up. Multiplicity adjustment for secondary outcome analyses |
| eTable 6 | A table showing the observed p values for all the secondary outcomes and ordered from the lower until the higher and the corrected p values using a Holm–Bonferroni correction |
| .T.L. 7 | Sensitivity Analyses for the Primary Outcome |
| eTable 7 | A table showing the proposed sensitivity analyses for the primary outcome (count analysis, common effect test, average relative effect test and heterogeneity of treatment effect) |
| | Characteristics of the Intervention |
| | A, Line plot reporting the mean and 95% confidence interval of the driving pressure after intubation, after recruitment maneuver, during first and second hour of surgery and at |
| eFigure 1 | the last hour by treatment group. B, Bar plot reporting the mean difference in driving pressure between groups after intubation, after recruitment maneuver, during first and second hour of surgery and at the last |
| Crigare r | hour. |
| | C, Bar plot showing the titrated level of PEEP in the individualized high PEEP group. |
| | D, Line plot showing the plateau pressure and driving pressure according to PEEP levels during the PEEP titration maneuver in the individualized high PEEP. |
| eFigure 2 | Level of PEEP in the Study Population |
| 3. 3. | Histogram reporting the most used level of PEEP during the first five hours of the surgical procedure by treatment group. |
| eFigure 3 | Tidal Volume, PEEP, Peak Pressure, Plateau Pressure, FiO <sub>2</sub> and SpO <sub>2</sub> During Surgery Line graph reporting the mean and 95% confidence interval of the variables after intubation, after recruitment maneuver, during first and second hour of surgery and at the last |
| Crigare 5 | hour by treatment group. |
| oFiguro 4 | VAS Pain, Respiratory Rate, SpO <sub>2</sub> and Mean Arterial Pressure During the First Five Days of Follow-Up |
| eFigure 4 | Line graph reporting the mean and 95% confidence interval of the variables in the first five days of follow-up by treatment group. |
| eFigure 5 | Patient Status in the First Five Days of Follow-Up |

| | Transition plot showing the status of the patients in the first five days of follow-up. |
|---|---|
| eFigure 6 | Confidence Distribution for the Primary Outcome Confidence distribution of the estimated absolute difference of the primary outcome of Individualized High PEEP versus Low PEEP constructed using a normal approximation. A, The full confidence distribution of the estimated absolute difference, with the dashed vertical line indicating the median value and the area highlighted in tan indicating the 95% confidence interval. The orange area is related to an absolute difference greater than 0 (i.e., the intervention is associated with higher incidence of PPC vs standard care). The dotted line at an absolute difference of 0 indicates no treatment effect. The figure demonstrates that the confidence probability that Individualized High PEEP is associated with a reduced incidence of PPC (to any extent) compared with Low PEEP is XX.X%. B, The cumulative confidence distribution of the estimated absolute difference, with the y-axis corresponding to the confidence the absolute difference is less than or equal to the value on the x-axis. The blue-gray area indicates a beneficial intervention (i.e., absolute difference lower than 0). The dashed vertical line indicates the median. |
| eFigure 7 | Results of the Sensitivity Analyses for the Primary Outcome Forest plot reporting the results of all sensitivity analyses |

Table 3 (Table 1) – Baseline Characteristics of the Included Patients

| | Individualized High PEED | Low PEEP |
|---|---|---|
| | Individualized High PEEP<br>(n = XXX) | (n = XXX) |
| Age, years | (n zox) | (11 - 1000) |
| Age ≥ 65 years – no. (%) | | |
| Male gender – no. (%) | | |
| Weight, kilograms | | |
| Body mass index, kg/m <sup>2</sup> | | |
| Body mass index ≥ 30 kg/m <sup>2</sup> | | |
| ARISCAT score | | |
| ARISCAT ≥ 45 – no. (%) | | |
| ASA physical status– no. (%) | | |
| 1 | | |
| 2 | | |
| 3 | | |
| 4 | | |
| Functional status – no. (%) | | |
| Independent | | |
| Partially dependent | | |
| Totally dependent | | |
| Co-existing disorders – no. (%) | | |
| Diabetes | | |
| Coronary artery disease | | |
| COPD | | |
| Smoker | | |
| Never | | |
| Former* | | |
| Current | | |
| Active cancer | | |
| Type of surgery – no. (%) | | |
| Urgent | | |
| Elective | | |
| Procedure – no. (%)** | | |
| Gynecology | | |
| Urology | | |
| Vascular | | |
| Pancreatic | | |
| Bowel | | |
| Liver | | |
| Gastric | | |
| Hepatic | | |
| Biliary | | |
| Other | | |
| Preoperative vital signs | | |
| Heart rate, bpm | | |
| · | | |

Table 3 (Table 1) – Baseline Characteristics of the Included Patients

| | Individualized High PEEP<br>(n = XXX) | Low PEEP<br>(n = XXX) |
|---|---|---|
| Systolic blood pressure, mmHg | | |
| Mean arterial pressure, mmHg | | |
| Respiratory rate, breaths/min | | |
| Temperature, °C | | |
| SpO <sub>2</sub> , % | | |
| $SpO_2 < 96\%$ - no. (%) | | |
| Preoperative chest X-ray – no. (%) | | |
| Infiltrates | | |
| Pleural effusion | | |
| Atelectasis | | |
| Preoperative laboratory | | |
| Hemoglobin, g/dL | | |
| Creatinine, mg/dL | | |

Data are median (quartile 25th - quartile 75th) or N / total (%).

Abbreviations: PEEP is positive end-expiratory pressure; ARISCAT is The Assess Respiratory Risk in Surgical Patients in Catalonia; ASA is American Society of Anesthesiology; COPD is chronic obstructive pulmonary disease;  $SpO_2$  is pulse oximetry.

<sup>\*</sup> Cessation more than 3 months.

<sup>\*\*</sup> A patient can have more than one.

Individualized

**High PEEP** 

(n = XXX)

**Low PEEP** 

(n = XXX)

**Absolute Difference** 

(95% CI)

p value

# Table 4 (Table 2) - Ventilation and Intraoperative Characteristics

| Table 4 (Table 2) – Ventilation and |
|----------------------------------------|
| Recruitment maneuver – no. (%) |
| Number of recruitment maneuvers |
| Lowest ΔP during PEEP titration, cmH2O |
| Tidal volume, mL/kg PBW |
| After intubation |
| During first hour |
| Last hour |
| PEEP, cmH <sub>2</sub> O |
| After intubation |
| During first hour |
| Last hour |
| Peak pressure, cmH <sub>2</sub> O |
| After intubation |
| During first hour |
| Last hour |
| Plateau pressure, cmH <sub>2</sub> O |
| After intubation |
| During first hour |
| Last hour |
| Driving pressure, cmH <sub>2</sub> O |
| After intubation |
| During first hour |
| Last hour |
| Respiratory rate, breaths/min |
| After intubation |
| During first hour |
| Last hour |
| FiO <sub>2</sub> |
| After intubation |
| During first hour |
| Last hour |
| SpO <sub>2</sub> , % |
| After intubation |
| During first hour |
| Last hour |
| etCO <sub>2</sub> , mmHg |
| After intubation |
| During first hour |

Last hour

#### Table 4 (Table 2) – Ventilation and Intraoperative Characteristics

| (n = XXX) (n = XXX) Mean arterial pressure, mmHg After intubation During first hour Last hour Duration of anesthesia, min Duration of surgery, min Duration of surgery ≥ 180 min – no. (%) Maintenance of anesthesia – no. (%) Volatile Totally intravenous anesthesia | <u> </u> | Individualized<br>High PEEP | Low PEEP<br>(n = XXX) | Absolute Difference<br>(95% CI) | p value |
|---|---|---|---|---|---|
| After intubation During first hour Last hour Duration of anesthesia, min Duration of surgery, min Duration of surgery ≥ 180 min – no. (%) Maintenance of anesthesia – no. (%) Volatile | <u>-</u> | (n = XXX) | (11 – XXX) | (93 // 01) | |
| During first hour Last hour Duration of anesthesia, min Duration of surgery, min Duration of surgery ≥ 180 min – no. (%) Maintenance of anesthesia – no. (%) Volatile | · | | | | |
| Last hour Duration of anesthesia, min Duration of surgery, min Duration of surgery ≥ 180 min – no. (%) Maintenance of anesthesia – no. (%) Volatile | | | | | |
| Duration of anesthesia, min Duration of surgery, min Duration of surgery ≥ 180 min – no. (%) Maintenance of anesthesia – no. (%) Volatile | | | | | |
| Duration of surgery, min Duration of surgery ≥ 180 min – no. (%) Maintenance of anesthesia – no. (%) Volatile | | | | | |
| Duration of surgery ≥ 180 min – no. (%) Maintenance of anesthesia – no. (%) Volatile | Duration of anesthesia, min | | | | |
| Maintenance of anesthesia – no. (%) Volatile | Duration of surgery, min | | | | |
| Volatile | Duration of surgery ≥ 180 min – no. (%) | | | | |
| | Maintenance of anesthesia – no. (%) | | | | |
| Totally intravenous anesthesia | Volatile | | | | |
| | Totally intravenous anesthesia | | | | |
| Combine | Combine | | | | |
| Epidural – no. (%) | Epidural – no. (%) | | | | |
| Thoracic | Thoracic | | | | |
| Lumbar | Lumbar | | | | |
| Neuromuscular monitoring – no. (%) | Neuromuscular monitoring - no. (%) | | | | |
| Residual paralysis at extubation– no. (%) | Residual paralysis at extubation– no. (%) | | | | |
| Paralysis reverted – no. (%) | Paralysis reverted – no. (%) | | | | |
| Temperature at the end of the surgery, °C | Temperature at the end of the surgery, °C | | | | |
| Fluids | Fluids | | | | |
| Total intake, mL | Total intake, mL | | | | |
| Crystalloids intake, mL | Crystalloids intake, mL | | | | |
| Colloid – no. (%) | Colloid – no. (%) | | | | |
| Colloid intake, mL | Colloid intake, mL | | | | |
| Total output, mL | Total output, mL | | | | |
| Urine output, mL | Urine output, mL | | | | |
| Blood loss, mL | Blood loss, mL | | | | |
| Fluid balance, mL | Fluid balance, mL | | | | |
| Transfusion – no. (%) | Transfusion – no. (%) | | | | |
| Packed red blood cells | Packed red blood cells | | | | |
| Fresh frozen plasma | Fresh frozen plasma | | | | |
| Platelets | Platelets | | | | |
| Unplanned ICU/HDU admission – no. (%) | Unplanned ICU/HDU admission – no. (%) | | | | |

Data are median (quartile 25th - quartile 75th) or N / total (%).

Abbreviation:  $\Delta P$  is driving pressure, PEEP is positive end-expiratory pressure, PBW is predicted body weight, FiO<sub>2</sub> is inspired fraction of oxygen, SpO<sub>2</sub> is pulse oximetry, etCO<sub>2</sub> is end-tidal carbon dioxide, ICU is intensive care unit, HDU is high dependency unit.

# Table 5 (eTable 2) – Additional Intraoperative Characteristics

| Table 6 (Crable 2) Additional in | Individualized High PEEP (n = XXX) | Low PEEP<br>(n = XXX) | Absolute Difference<br>(95% CI) | p value |
|---|---|---|---|---|
| Fluids | | | | |
| Total intake, mL | | | | |
| Crystalloids – no. (%) | | | | |
| Cumulative intake, mL | | | | |
| Colloid – no. (%) | | | | |
| Cumulative intake, mL | | | | |
| Total output, mL | | | | |
| Urine output – no. (%) | | | | |
| Cumulative output, mL | | | | |
| Blood loss – no. (%) | | | | |
| Cumulative loses, mL | | | | |
| Fluid balance, mL | | | | |
| Vasopressors | | | | |
| Dobutamine – no. (%) | | | | |
| Cumulative dose, mg | | | | |
| Dopamine – no. (%) | | | | |
| Adrenaline – no. (%) | | | | |
| Cumulative dose, mg | | | | |
| Ephedrine – no. (%) | | | | |
| Cumulative dose, mg | | | | |
| Noradrenaline – no. (%) | | | | |
| Cumulative dose, mg | | | | |
| Phenylephrine – no. (%) | | | | |
| Cumulative dose, mg | | | | |
| Transfusion | | | | |
| Packed red blood cells – no. (%) | | | | |
| Cumulative amount, mL | | | | |
| Fresh frozen plasma – no. (%) | | | | |
| Cumulative amount, mL | | | | |
| Platelets – no. (%) | | | | |

Data are median (quartile 25th - quartile 75th) or N / total (%). Abbreviations: PEEP is positive end-expiratory pressure.

Cumulative amount, mL

Individualized

**High PEEP** 

(n = XXX)

**Low PEEP** 

(n = XXX)

**Absolute Difference** 

(95% CI)

p value

# Table 6 (eTable 3) – Daily Assessment of Included Patients

| Day 1 |
|-------------------------------------|
| Patients in hospital – no. (%) |
| Admission to ICU – no. (%) |
| Mechanical ventilation – no. (%) |
| Invasive |
| Non-invasive |
| Physiotherapy – no. (%) |
| Renal replacement therapy – no. (%) |
| VAS pain |
| Respiratory rate, breaths/min |
| SpO <sub>2</sub> , % |
| Mean arterial pressure, mmHg |
| Day 2 |
| Patients in hospital – no. (%) |
| Admission to ICU – no. (%) |
| Mechanical ventilation – no. (%) |
| Invasive |
| Non-invasive |
| Physiotherapy – no. (%) |
| Renal replacement therapy – no. (%) |
| VAS pain |
| Respiratory rate, breaths/min |
| SpO <sub>2</sub> , % |
| Mean arterial pressure, mmHg Day 3 |
| Patients in hospital – no. (%) |
| Admission to ICU – no. (%) |
| Mechanical ventilation – no. (%) |
| Invasive |
| Non-invasive |
| Physiotherapy – no. (%) |
| Renal replacement therapy – no. (%) |
| VAS pain |
| Respiratory rate, breaths/min |
| SpO <sub>2</sub> , % |
| Mean arterial pressure, mmHg |
| Day 4 |
| Patients in hospital – no. (%) |
| Admission to ICU – no. (%) |
| Mechanical ventilation – no. (%) |
| Invasive |

# Table 6 (eTable 3) - Daily Assessment of Included Patients

| | Individualized<br>High PEEP<br>(n = XXX) | Low PEEP (n = XXX) | Absolute Difference<br>(95% CI) | p value |
|---|---|---|---|---|
| Non-invasive | | | | |
| Physiotherapy – no. (%) | | | | |
| Renal replacement therapy – no. (%) | | | | |
| VAS pain | | | | |
| Respiratory rate, breaths/min | | | | |
| SpO <sub>2</sub> , % | | | | |
| Mean arterial pressure, mmHg | | | | |
| Day 5 | | | | |
| Patients in hospital – no. (%) | | | | |
| Admission to ICU – no. (%) | | | | |
| Mechanical ventilation – no. (%) | | | | |
| Invasive | | | | |
| Non-invasive | | | | |
| Physiotherapy – no. (%) | | | | |
| Renal replacement therapy – no. (%) | | | | |
| VAS pain | | | | |
| Respiratory rate, breaths/min | | | | |
| SpO <sub>2</sub> , % | | | | |
| Mean arterial pressure, mmHg | | | | |

Data are median (quartile 25th - quartile 75th) or N / total (%).

Abbreviations: PEEP is positive end-expiratory pressure, ICU is intensive care unit, VAS is visual analogue scale, SpO<sub>2</sub> is pulse oximetry.

#### Table 7 (Table 3) – Primary and Secondary outcomes

| Individualized High PEEP $(n = XXX)$ Low Pingle ( $n = X$ ) | p value |
|-------------------------------------------------------------|---------|
|-------------------------------------------------------------|---------|

#### **Primary outcome**

Postoperative pulmonary complications - no. (%)

Severe respiratory failure

Bronchospasm

Suspected pulmonary infection

Pulmonary infiltrates

Aspiration pneumonitis

Atelectasis

Acute respiratory distress syndrome

Pleural effusion

Cardiopulmonary edema

Pneumothorax

#### **Secondary outcomes**

Mild respiratory failure - no. (%)

Intraoperative complications – no. (%)

Desaturation

Hypotension

Need for vasoactive agents

New arrhythmias

Postoperative extrapulmonary complications – no. (%)

Sepsis

Septic shock

Extrapulmonary infection

Anastomotic leakage

Acute kidney injury

Intraoperative fluid balance - no. (%)

Impaired wound healing – no. (%)

Unplanned admission to intensive care unit – no. (%)

Intensive care unit length of stay, days

Hospital length of stay, days

All-cause hospital mortality - no. (%)

Data are median (quartile 25th - quartile 75th) or N / total (%). Abbreviations: PEEP is positive end-expiratory pressure.

# **MODIFICATIONS FROM THE ORIGINAL ANALYSIS PLAN**

| ANALYSIS | ORIGINAL PLAN<br>( <i>TRIALS</i> 2020; 21:198) | UPDATE IN THE SAP<br>(Closed in January 12, 2024) | INCLUDED IN THE NEW SAP (Updated in January 12, 2025) |
|---|---|---|---|
| Model for the primary outcome | Risk ratio and 95% confidence intervals calculated with Wald's likelihood ratio approximation test and with $\chi^2$ tests for hypothesis testing. | Mixed-effect generalized linear model with binomial distribution and identity link, with sites included as random effects to account for the clustering effect and reported as absolute difference with a two–sided 95% confidence interval. | |
| Model for binary secondary outcomes | Risk ratio and 95% confidence intervals calculated with Wald's likelihood ratio approximation test and with $\chi^2$ tests for hypothesis testing. | Mixed-effect generalized linear model with binomial distribution and identity link, with sites included as random effects to account for the clustering effect and reported as absolute difference with a two–sided 95% confidence interval. | |
| Model for ICU and hospital length of stay | Generalized linear models considering distributions that will fit a possible heavy right-tailed distribution without zero (such as truncated Poisson, gamma distribution, or inverse Gaussian), choosing the best fit according to the model's deviance. | Mixed-effect median regression with sites also including as clustering effect, and reported as median difference with a two–sided 95% confidence interval. | |
| Time-to-event<br>analyses | Kaplan–Meier curves will be used to report time to postoperative pulmonary complications, and hazard ratios with a 95% confidence interval will be calculated with Cox proportional hazard models without adjustment for covariates. | No time-to-event analysis planned to be performed. | |
| Subgroup analysis | Analyses of heterogeneity of effects across subgroups will be performed with the use of treatment-by-subgroup interaction term, added to a generalized linear model considering a binomial distribution, and will be presented in a forest plot. | Analyses of heterogeneity of effects across subgroups will be performed with the use of treatment-by-subgroup term added to the primary model and will be presented in a forest plot. | |
| Additional analyses | Not described. | Since the primary outcome of the present study is a composite one, the choice of the statistical method is an important part of designing because various methods | |

| | | provide different power, depending on the situation. In addition to the standard analysis described above, additional analyses will be performed. | |
|---|---|---|---|
| Confidence<br>distribution | Not described. | Not described. | To support interpretation, a confidence distribution for the primary outcome using a normal approximation on the estimated absolute difference will be calculated. The confidence distribution will be computed to provide the frequentist probability that the absolute difference is less than 0.10 In addition, the confidence distribution will be reported in a plot. |

Abbreviations: ICU: intensive care unit.

#### **PROPOSED FIGURE 1**

